CLINICAL TRIAL: NCT00449007
Title: A Randomized Controlled Study Comparing Fluoxetine With Bupropion for Impulsivity and Suicidality in Patients With Major Depressive Disorder and Comorbid Alcoholism (Abuse or Dependence)
Brief Title: Fluoxetine and Bupropion to Treat Patients With Depression and Alcoholism
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment of this population was not feasible
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAA-OQU-015630-02; P20AA015630 (NIH); NIH Grant P20 AA015630-02
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Depression; Alcoholism; Suicidal Behavior
Keywords: Major depressive disorder; Alcohol abuse; Alcohol dependence; Suicide
MeSH Terms: conditions — Depression; Alcoholism; Depressive Disorder, Major; Suicide | interventions — Fluoxetine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): fluoxetine -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  Interventions: Drug: fluoxetine
- 2 (Active Comparator): bupropion -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  Interventions: Drug: bupropion

INTERVENTIONS:
Drug: fluoxetine — 6 months
  Arms: 1
Drug: bupropion — 6 months
  Arms: 2

SUMMARY:
We will study patients with a current major depressive episode, comorbid alcoholism and a history of a past suicide attempt. All subjects with alcohol dependence will be evaluated for risk of alcohol withdrawal prior to randomization. The study will provide six months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention. Patients will also be encouraged to attend daily Alcoholics Anonymous meetings. The outcome measures will be: 1) occurrence of suicide events; 2) reduction of suicidal ideation; 3) reduction in neuropsychological measures of impulsivity.

DETAILED DESCRIPTION:
Suicide is a significant public health problem. Depression, alcoholism (abuse or dependence), and a prior suicide attempt are risk factors for suicide. However, little information exists to guide clinicians in the choice of antidepressant medication for patients with comorbid major depression and alcoholism who are at risk for suicidal acts.

There is evidence that selective serotonin reuptake inhibitors (SSRI) may reduce impulsive aggression, and therefore lower the risk for suicidal behavior. We will test the hypothesis that fluoxetine, an SSRI, will be associated with fewer suicide events (defined as suicidal acts or increases in suicidal ideation necessitating a change in management), decreased suicidal ideation and decreases in neuropsychological measures of impulsivity compared to bupropion. The non-serotonergic drug, bupropion will improve energy and hopelessness. We expect the two drugs to be equally efficacious in reducing global depression severity. We will compare fluoxetine with bupropion in a 6-month randomized, controlled study of major depressive disorder and comorbid alcoholism in patients who have a prior history of suicide attempt. Patients requiring alcohol detoxification will be excluded. Patients will also receive weekly psychotherapy.

We will study 42 subjects with a current major depressive episode, comorbid alcoholism and a history of a past suicide attempt (21 subjects per year) in a randomized, double-blind, controlled trial, stratified by alcoholism type (1 vs 2). All subjects with alcohol dependence will be evaluated for risk of alcohol withdrawal prior to randomization. We will include patients who have suicidal ideation. However, patients with a suicidal plan or intent will only be enrolled as inpatients if the research team and the independent treatment team on the inpatient research unit agree that this is clinically reasonable. For example, if ECT or antipsychotics are indicated, the patient will not be enrolled. The study will provide six months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention. Patients will also be encouraged to attend daily Alcoholics Anonymous meetings. The outcome measures will be: 1) occurrence of suicide events; 2) reduction of suicidal ideation; 3) reduction in neuropsychological measures of impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a major depressive episode (unipolar only) AND alcohol dependence or abuse; Score of greater than 16 on the HDRS
* Age range 18-65 years
* History of a past suicide attempt, defined as self destructive behavior with at least some intent to die; patients with suicidal plan or intent will only be enrolled as inpatients if staff agrees it is reasonable.
* Able to tolerate cross taper to study medications

Exclusion Criteria:

* Other major psychiatric disorders such as Bipolar Disorder; schizophrenia or schizoaffective disorder, past or current psychotic symptoms; eating disorder; substance abuse or dependence (other than alcohol, caffeine or nicotine); persons already taking SSRIs or bupropion for other indications such as anxiety disorders.
* Primary disorder is an anxiety disorder such as Panic disorder/GAD/OCD/Social anxiety disorder, with secondary depression.
* CIWA-AR rating >10 or history of delirium tremens or seizures.
* Blood pressure >150 systolic or >90 diastolic
* Active or untreated medical problems
* Antipsychotic medication required
* History of becoming hypomanic or manic on antidepressants
* Contraindication to the use of fluoxetine or bupropion, or currently using Zyban
* Failure to respond to adequate trials of 3 SSRIs or fluoxetine or bupropion in the last 2 years (failure to respond to therapeutic trial defined as: at least 2/3 maximal PDR dose for at least 6 weeks)
* Lack of capacity to consent
* Pregnancy, lactation, or plans to conceive during the course of study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Oquendo, MD, Principal Investigator — NYS Psychiatric Institute / Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine: fluoxetine -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  fluoxetine: 6 months
- Bupropion: bupropion -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  bupropion: 6 months
Period: Overall Study
Arm/Group | Fluoxetine | Bupropion
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Bupropion | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (3.8) | 33.5 (10.6) | 37.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Suicide Events Either a Suicide Death, a Suicide Attempt, or Suicidal Ideation Severe Enough to Warrant a Medical Intervention
Description: patients have either a suicide death, a suicide attempt, or suicidal ideation severe enough to warrant a medical intervention. this is assessed using the Columbia Suicide History Form and a consensus conference rules on whether the event meets criteria or not. Medical interventions can include hospitalization, a change in medication (adding adjunctive meds) or an increase in frequency of visits or other methods to monitor the patient.
  The range is 0 and up and denotes the number of suicide events (not the number of participants and not the number of suicide attempts). Higher score is worse and predicts future suicidal behavior
Time Frame: 6 months
Population: patients randomized to one of two arms for 6 months and assessed weekly for 8 weeks and then monthly
Measure: Number; unit: suicide events
Groups:
- Fluoxetine for 6 Months: fluoxetine -- patients randomized to one of two arms for 6 months and assessed weekly for 8 weeks and then monthly. patients receive 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  fluoxetine: 6 months
- Bupropion for 6 Months: bupropion fluoxetine -- patients randomized to one of two arms for 6 months and assessed weekly for 8 weeks and then monthly. patients receive 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  : bupropion: 6 months
Arm/Group | Fluoxetine for 6 Months | Bupropion for 6 Months
Number analyzed (Participants) | 2 | 3
suicide events | 2 | 3

2. Secondary Outcome: Suicidal Ideation at 6 Months
Description: Participant Score on the Scale for Suicidal Ideation will be the outcome variable.
  The SSI range is from 0-38 and higher score is worse and may predict suicide risk
Time Frame: 6 month
Population: All 5 participants had data and calculated scores for the Scale for Suicidal Ideation during the conduct of the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluoxetine 6 Months of Antidepressant: fluoxetine -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  fluoxetine: 6 months
- Bupropion 6 Months of Antidepressant: bupropion -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  bupropion: 6 months
Arm/Group | Fluoxetine 6 Months of Antidepressant | Bupropion 6 Months of Antidepressant
Number analyzed (Participants) | 2 | 3
units on a scale | 0.5 (0.7) | 8.5 (12.0)
Statistical Analysis 1: Comparison: Bupropion 6 Months of Antidepressant; Difference between 6 months and baseline for Bupropion treated group. Due to the low number of participants, the results are unreliable; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4.5

ADVERSE EVENTS:
Groups:
- Arm 1 Randomized to Fluoxetine: fluoxetine -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  fluoxetine: 6 months
- Arm 2 Randomized to Bupropion: bupropion -- 6 months of antidepressant pharmacotherapy as well as psychotherapy focused on alcohol relapse prevention; patients will also be encouraged to attend daily Alcoholics Anonymous meetings
  bupropion: 6 months
Arm/Group | Arm 1 Randomized to Fluoxetine | Arm 2 Randomized to Bupropion
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No